CLINICAL TRIAL: NCT04900896
Title: Outcome Measures Study on an Adult Myoelectric Elbow-Wrist-Hand Orthosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Myomo (Industry)
Collaborators: Orthocare Innovations, LLC (Industry); Geauga Rehabilitation Engineering, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRO-001
Record Dates: First submitted 2021-05-12; First posted 2021-05-25 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Brachial Plexus Injury; Spinal Cord Injuries; Neurological Disease
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Myoelectric Elbow-Wrist-Hand Orthosis — An arm orthosis that uses myoelectric signals to control the level of mechanical assistance provided to a user's elbow and hand in order to overcome upper limb weakness or paralysis and achieve functional tasks.
  Other Names: MyoPro®

SUMMARY:
The objective of this study is to evaluate the therapeutic and functional gains of a myoelectric elbow-wrist-hand orthosis for adult individuals with upper limb impairments using repeated measures studies that combines both gross motion and quantitative function outcome measures.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the therapeutic and functional gains of a myoelectric elbow-wrist-hand orthosis for adult individuals with upper limb impairments using repeated measures studies that combines both gross motion and quantitative function outcome measures.

The primary outcomes of this study will collect data on the participants' therapeutic and functional outcome measures when using the MyoPro over time in their home. Baseline data without the device will be collected prior to receiving the MyoPro. Data with and without the device will then be collected at 2-weeks post fitting and then at 1-month intervals thereafter for 12 months. These outcome measures will enable an understanding of the participants' functional gains with and without the MyoPro and over time with the MyoPro.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years and older
* Upper limb impairment caused by brachial plexus injury (BPI), any stroke (CVA), spinal cord injury (SCI), or other neurological diagnoses
* Be medically stable
* Be in the process of being fit with a MyoPro as a first-time user
* Has at least trace muscle activation in the elbow and wrist flexors and extensors as measured by a 1/5 on a manual muscle test at targeted joints
* Has the minimum microvolt EMG threshold to operate the MyoPro, such that the individual can sustain the EMG signals above the threshold for two full seconds (both at elbow and hand) for a minimum of three times within three minutes
* Has passive range of motion within 5 degrees of terminal range for finger open and close
* Has passive range of motion within 5 degrees of terminal range for wrist flexion and at least neutral for wrist extension
* Has passive range of motion within 5 degrees of terminal range for elbow flexion and extension
* Has at least 30 degrees of active range of motion for shoulder flexion or shoulder abduction
* Able to support the weight of the MyoPro
* Able to tolerate functional tasks for 20 min with intermittent rests without excessive fatigue
* Has intact cognition
* Able to clearly and verbally communicate in the English language
* Has a wireless internet connection to participate in telehealth sessions
* Be attending therapy within four weeks of getting fit and trained with a MyoPro

Exclusion Criteria:

* Has a body weight above 235 lbs
* Upper limb measurements will not allow for correct fit of the orthosis.
* Fixed upper limb contractures on affected side
* Unable to have full passive finger opening when the wrist is in neutral
* Severe spasticity or tone defined as 2 or higher at the wrist or fingers, or 3 or higher at the elbow on the Modified Ashworth Spasticity Scale
* Severe shoulder subluxation (greater than one finger with significant pain) or shoulder dislocation
* Passive shoulder range of motion less than 45 degrees in flexion and abduction
* Excessive pain, hypersensitivity, or skin issues in the arm(s) that would prevent wearing the MyoPro
* Severe cognitive or psychiatric problems that might be contraindicated for training and safe MyoPro use
* Bilateral upper limb impairment
* Pregnancy
* Other conditions (e.g. history of neurological disorder other than SCI, BPI, or CVA) or circumstances that would preclude safe and/or effective participation, including severe sensory deficits, skin conditions, and/or other sequelae that may be contraindicated for myoelectric MyoPro use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with upper limb impairment caused by brachial plexus injury, stroke, or spinal cord injury, or other neurological disease or injury who have no fixed upper limb contractures on the affected side and have been fitted with a myoelectric Elbow-Wrist-Hand orthosis.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to after intervention in Shoulder Flexion Strength | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  A manual muscle test (MMT) will be conducted to measure shoulder flexion strength of the affected arm.
Change from baseline to after intervention in Shoulder Abduction Strength | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  A manual muscle test (MMT) will be conducted to measure shoulder abduction strength of the affected arm.
Change from baseline to after intervention in Bicep Strength | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  A manual muscle test (MMT) will be conducted to measure bicep strength of the affected arm.
Change from baseline to after intervention in Triceps Strength | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  A manual muscle test (MMT) will be conducted to measure triceps strength of the affected arm.
Change from baseline to after intervention in Hand Grip Strength | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  A manual muscle test (MMT) or dynamometer will be used to measure hand grip strength of the affected arm.
Change from baseline to after intervention in Modified Ashworth Scale: Bicep | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Bicep muscle spasticity of the affected arm will be measured according to the Modified Ashworth Scale.
Change from baseline to after intervention in Modified Ashworth Scale: Triceps | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Triceps muscle spasticity of the affected arm will be measured according to the Modified Ashworth Scale.
Change from baseline to after intervention in Modified Ashworth Scale: Wrist Flexors | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Wrist flexors muscle spasticity of the affected arm will be measured according to the Modified Ashworth Scale.
Change from baseline to after intervention in Modified Ashworth Scale: Wrist Extensors | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Wrist extensors muscle spasticity of the affected arm will be measured according to the Modified Ashworth Scale.
Change from baseline to after intervention in Modified Ashworth Scale: Finger Flexors | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Finger flexors muscle spasticity of the affected arm will be measured according to the Modified Ashworth Scale.
Change from baseline to after intervention in Modified Ashworth Scale: Finger Extensors | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Finger extensors muscle spasticity of the affected arm will be measured according to the Modified Ashworth Scale.
Change from baseline to after intervention in Active Range of Motion: Shoulder Flexion | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active shoulder flexion range of motion of the affected arm will be measured.
Change from baseline to after intervention in Active Range of Motion: Shoulder Extension | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active shoulder extension range of motion of the affected arm will be measured.
Change from baseline to after intervention in Active Range of Motion: Shoulder Abduction | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active shoulder abduction range of motion of the affected arm will be measured.
Change from baseline to after intervention in Active Range of Motion: Shoulder Adduction | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active shoulder adduction range of motion of the affected arm will be measured.
Change from baseline to after intervention in Active Range of Motion: Elbow Flexion | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active elbow flexion range of motion of the affected arm will be measured.
Change from baseline to after intervention in Active Range of Motion: Elbow Extension | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active elbow extension range of motion of the affected arm will be measured.
Change from baseline to after intervention in Active Range of Motion: Wrist Flexion | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active wrist flexion range of motion of the affected arm will be measured.
Change from baseline to after intervention in Active Range of Motion: Wrist Extension | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Active wrist extension range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Shoulder Flexion | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive shoulder flexion range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Shoulder Extension | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive shoulder extension range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Shoulder Abduction | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive shoulder abduction range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Shoulder Adduction | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive shoulder adduction range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Elbow Flexion | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive elbow flexion range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Elbow Extension | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive elbow extension range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Wrist Flexion | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive wrist flexion range of motion of the affected arm will be measured.
Change from baseline to after intervention in Passive Range of Motion: Wrist Extension | Once at baseline; once after intervention at midway through therapy (anticipated at 4 weeks); once after intervention at discharge from therapy (anticipated at 8 weeks)
  Passive wrist extension range of motion of the affected arm will be measured.
Functional Timed Tasks Score | Baseline, 2-weeks post fitting, monthly for 12-months post fitting
  Participants will complete a pre-identified battery of functional timed tasks that will be scored.
Functional Timed Tasks Time | Baseline, 2-weeks post fitting, monthly for 12-months post fitting
  Participants will complete a pre-identified battery of functional timed tasks that will be timed.

SECONDARY OUTCOMES:
Elbow flex/extend | 2-weeks post fitting, monthly for 12-months post fitting
  The number of elbow flex/extend repetitions per day will be recorded.
Hand open/close | 2-weeks post fitting, monthly for 12-months post fitting
  The number of hand open/close repetitions per day will be recorded.
Quality of life rating | Baseline, 2-weeks post fitting, monthly for 12-months post fitting
  Participants will be asked to rate their quality of life from "Very Poor" to "Very Good".

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Chang, PhD, Principal Investigator — Orthocare Innovations, LLC
Locations (3):
- United States (3):
  - Myomo, Inc., Boston, Massachusetts
  - Geauga Rehabilitation Engineering, Inc., Chardon, Ohio
  - Orthocare Innovations, LLC, Edmonds, Washington

IPD SHARING:
Plan to Share IPD: No